CLINICAL TRIAL: NCT02783521
Title: Feasibility of a Gender- and Culturally-Sensitive Weight Loss Intervention for Hispanic Males
Brief Title: Gender- and Culturally-Sensitive Weight Loss Intervention for Hispanic Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1604536275
Record Dates: First submitted 2016-05-20; First posted 2016-05-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Overweight; Obesity
Keywords: Hispanic men; Weight loss; Diet; Physical activity; Intervention
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Includes changing eating behaviors, increasing physical activity, and attending regular in-person weight loss meetings for 12 weeks. To support additional weight loss/weight maintenance, participants will receive bi-weekly phone calls across a 12 week follow-up.
  Interventions: Behavioral: Counseling sessions
- Wait List Control (Other): Wait-list control participants will not receive any intervention for the first 12 weeks. After 12 weeks, participants will receive the weight loss intervention plus mHealth technology support.
  Interventions: Behavioral: Wait List Control

INTERVENTIONS:
Behavioral: Counseling sessions — During the first 12 weeks, intervention participants will attend weekly 30-45-minute individual counseling sessions guided by a trained bilingual Hispanic male lifestyle coach. Counseling sessions will be tailored to the needs of the participants (e.g., evening/weekend sessions, waiting/childcare area). After 12 weeks, intervention group participants will receive bi-weekly phone calls across a 12-week follow-up. Phone calls will last approximately 10 minutes in duration and study staff will follow a script to review current body weight, eating and activity behaviors, and specific barriers for weight loss/maintenance or diet/physical activity behaviors.
  Arms: Intervention
Behavioral: Wait List Control — After 12 weeks, the wait list control will receive the weight loss intervention plus mHealth technology support. It will include tailored, targeted text messaging and real-time self-monitoring support including beverage tracking cups, which provide the amount of calories users are consuming through beverages on a daily basis, and wearable activity monitors.Behavioral constructs used for the intervention group will be maintained during this intervention delivery thereby ensuring all participants have the appropriate tools to continue weight loss efforts regardless of mHealth use.
  Arms: Wait List Control

SUMMARY:
The investigators propose to 1) assess the feasibility, acceptability and preliminary efficacy of a gender- and culturally-sensitive weight loss intervention in 48 overweight/obese Hispanic males ages 18-64 over 12 weeks; 2) assess participant characteristics and process measures related to the uptake of mobile-health (mHealth) technology in overweight/obese Hispanic males over 12 weeks; and 3) assess pathologic changes in the liver in Hispanic men enrolled in a 12-week weight loss intervention using a non-invasive MRI as a therapeutic response biomarker.

DETAILED DESCRIPTION:
In the U.S., Hispanic males have the highest rate of overweight and obesity when compared to males of other racial/ethnic groups placing them at greater risk for obesity-related disease. Yet, current literature is lacking to inform on best practices to engage Hispanic males in weight loss and/or to promote a successful weight loss trajectory. Without this information the health disparities associated with obesity and obesity-related chronic disease will continue. Evidence exists to support behavioral weight loss in reducing obesity-related health risks. There are limited data to suggest these programs are effective for men and no data to support the feasibility and effectiveness of these programs among Hispanic males despite this being the fastest growing and highest burdened group for obesity-related disease within the U.S. population. Using existing practice guidelines and evidence from recently completed in-depth qualitative interviews in overweight/obese Hispanic males, the investigators will test a novel intervention approach to address this gap in knowledge. The investigators propose to 1) assess the feasibility, acceptability and preliminary efficacy of a gender- and culturally-sensitive weight loss intervention in 48 overweight/obese Hispanic males ages 18-64 over 12 weeks; 2) assess participant characteristics and process measures related to the uptake of mobile-health (mHealth) technology in overweight/obese Hispanic males over 12 weeks; and 3) assess pathologic changes in the liver in Hispanic men enrolled in a 12-week weight loss intervention using a non-invasive MRI as a therapeutic response biomarker. This project will challenge current research paradigms for Hispanic males by testing a gender- and culturally-sensitive weight loss intervention and providing highly impactful formative research on the use of novel mHealth self-monitoring technologies to facilitate dietary/physical activity behavior changes. Given the Hispanic population is the fastest growing in the U.S., efforts to identify strategies to promote weight control among Hispanic males has potential to significantly impact public health. The expected outcome of the proposed project is the identification of feasible and appropriate weight loss intervention strategies to improve engagement and weight management in this vulnerable ethnic group.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* BMI between 25 to 45.0 kg/m² (NOTE: The investigators elected to cap this at 45.0 kg/m² to minimize potential risks and to reduce the potential for obesity to limit exercise participation)
* Ability to provide informed consent and health risk assessment prior to participation in this study
* Speak, read, and write either English and/or Spanish

Exclusion Criteria:

* Uncontrolled diabetes mellitus
* History of bariatric surgery
* Report medical condition or treatment for a medical condition that could affect body weight or ability to engage in structured physical activity that is consistent with the intervention for this study
* Current congestive heart failure, angina, uncontrolled arrhythmia, or other symptoms indicative of an increased acute risk for a cardiovascular event
* Resting systolic blood pressure of ≥150 mmHg or resting diastolic blood pressure of ≥90 mmHg
* Eating disorders that would contraindicate weight loss or physical activity
* Alcohol or substance abuse
* Currently treated for psychological issues (i.e. depression, bipolar disorder, etc.), taking psychotropic medications with the previous 12 months, or hospitalized for depression within the previous 5 years
* Report exercise on ≥3 days per week for ≥ 20 minutes per day over the past 3 months
* Report weight loss of ≥5% or participating in a weight reduction diet program in the past 3 months
* Report plans to relocate to a location that limits their access to the study site or having employment, personal, or travel commitments that prohibit attendance to all of the scheduled assessments

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Study Recruitment: Interest in Participation | Baseline
  The number of Hispanic men who contact the researchers and express interest in participation.
Study Recruitment: Screened for Eligibility | Baseline
  The number of Hispanic men screened for eligibility.
Study Recruitment: Eligibility | Baseline
  The number of Hispanic men eligible/ineligible for study inclusion and reason for ineligibility.
Study Recruitment: Enrollment | Baseline
  The number of Hispanic men enrolled in the study.
Retention | Week 24
  Retention will be measured as the number of participants who remain in the study at 24 weeks, divided by the number enrolled.
Treatment Satisfaction/Acceptability | Week 24
  Participants will be asked to rate their overall satisfaction with the intervention at 24 weeks and if they would recommend the program to others. Participants will also be asked questions regarding satisfaction with their overall progress and for changing dietary and PA habits, and weight

SECONDARY OUTCOMES:
Change in body weight. | 6, 12, 18, and 24 weeks
  Body weight will be measured on a digital scale to assess change in body weight over the intervention period.
Change in physical activity | 6, 12, 18, and 24 weeks
  A questionnaire will be used to measure and quantify energy expenditure from physical activity.
Change in dietary intake | 12 and 24 weeks
  A questionnaire will be used to assess self-reported food intake. This will be used to estimate calories, dietary fat, protein, and carbohydrates used.
Change in liver fat content (intervention only) | 12 weeks
  A non-invasive MRI will be used to assess changes in liver fat content for intervention participants at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: David O. Garcia, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Collaboratory for Metabolic Disease Prevention and Treatment, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Lindberg NM, Stevens VJ, Halperin RO. Weight-loss interventions for Hispanic populations: the role of culture. J Obes. 2013;2013:542736. doi: 10.1155/2013/542736. Epub 2013 Feb 26. PMID 23533725
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Pagoto SL, Schneider KL, Oleski JL, Luciani JM, Bodenlos JS, Whited MC. Male inclusion in randomized controlled trials of lifestyle weight loss interventions. Obesity (Silver Spring). 2012 Jun;20(6):1234-9. doi: 10.1038/oby.2011.140. Epub 2011 Jun 2. PMID 21633403
- [Background] Garcia DO, Valdez LA, Hooker SP. Hispanic Male's Perspectives of Health Behaviors Related to Weight Management. Am J Mens Health. 2017 Sep;11(5):1547-1559. doi: 10.1177/1557988315619470. Epub 2015 Dec 3. PMID 26634854
- [Derived] Garcia DO, Valdez LA, Aceves B, Bell ML, Rabe BA, Villavicencio EA, Marrero DG, Melton F, Hooker SP. mHealth-Supported Gender- and Culturally Sensitive Weight Loss Intervention for Hispanic Men With Overweight and Obesity: Single-Arm Pilot Study. JMIR Form Res. 2022 Sep 21;6(9):e37637. doi: 10.2196/37637. PMID 36129735
- [Derived] Garcia DO, Valdez LA, Bell ML, Humphrey K, Hingle M, McEwen M, Hooker SP. A gender- and culturally-sensitive weight loss intervention for Hispanic males: The ANIMO randomized controlled trial pilot study protocol and recruitment methods. Contemp Clin Trials Commun. 2018 Feb 9;9:151-163. doi: 10.1016/j.conctc.2018.01.010. eCollection 2018 Mar. PMID 29696238